CLINICAL TRIAL: NCT01362985
Title: Monitoring of Plerixafor Off-Label Use in the European Group for Blood and Bone Marrow Transplantation (EBMT) Registry
Brief Title: Analysis of Data Collected in the European Group for Blood and Marrow Transplantation (EBMT) Registry for Off-Label Transplant Use of Plerixafor
Status: Completed | Type: Observational
Sponsor: Genzyme, a Sanofi Company (Industry)
Collaborators: European Society for Blood and Marrow Transplantation (Network)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: MOZ19310; OBS13612 (Other: Sanofi)
Record Dates: First submitted 2011-05-27; First posted 2011-06-01 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Acute Leukemia; Chronic Leukemia; Myelodysplastic Syndrome; Myeloproliferative Neoplasm; Solid Tumors; Lymphoma; Plasma Cell Disorders
MeSH Terms: conditions — Myelodysplastic Syndromes; Myeloproliferative Disorders; Lymphoma

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

SUMMARY:
Genzyme will evaluate/monitor the off label transplant use of plerixafor using data in the European Group for Blood and Marrow Transplantation (EBMT) registry. Off-label use of plerixafor will be collected for data entered over a 5 year time span (i.e., data entered into the registry between the date of European Union (EU) marketing authorization [31 July 2009] and 31 July 2014).

The EBMT is a non-profit, scientific society representing more than 600 transplant centers mainly in Europe. The EBMT promotes all activity aiming to improve stem cell transplantation or cellular therapy, which includes registering all the activity relating to stem cell transplants. Data are entered, managed, and maintained in a central database with internet access; each EBMT center is represented in this database.

The collection by the EBMT registry of reasons for the off-label transplant use of plerixafor shall provide information of a substantial number of patients who are representative of the patient population receiving plerixafor off-label.

ELIGIBILITY:
Inclusion Criteria: Patients treated with plerixafor who have 1 or more of the following:

* Background disease other than lymphoma or multiple myeloma (MM)
* Are younger than 18 years of age.
* Received transplant using ex vivo plerixafor-mobilised cells (umbilical cord cell, peripheral blood (PB), bone marrow (BM) cell collection)
* Received treatment with plerixafor alone (i.e., without granulocyte colony stimulating factor (G-CSF))
* Contraindication for G-CSF
* Transplants using plerixafor-mobilised cells from allogeneic donor
* Received transplant using plerixafor-mobilised bone marrow cells
* Routes of plerixafor administration other than subcutaneous
* Patients whose cells do not mobilize poorly
* Other

Exclusion Criteria:

* Adults diagnosed with lymphoma or multiple myeloma (MM) and have been treated with plerixafor according to the European Union (EU) label.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients treated off-label with plerixafor.
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2009-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Number of patients who received plerixafor outside of the label indication in Europe and the reason for administration | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company